CLINICAL TRIAL: NCT02973776
Title: Vasoconstriction Trial Comparing LEO 90100 With Dermovate Cream, Diprosone Ointment, Elocon Cream, Locoid Ointment and LEO 90100 Vehicle
Brief Title: Vasoconstriction Trial With LEO 90100 Aerosol Foam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LP0053-1276
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — betamethasone-17,21-dipropionate; Mometasone Furoate; hydrocortisone-17-butyrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LEO 90100 aerosol foam (Experimental): LEO 90100 calcipotriol 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate) aerosol foam
  Each subject has all 6 treatments applied topically at the same time, however, the location on which the treatments are applied is randomised. Subjects will receive approximately 20 μl of each investigational product applied in circles with a diameter of 2.2 cm once.
  Interventions: Drug: LEO 90100 aerosol foam; Drug: Dermoval®/Dermovate®; Drug: Diprosone; Drug: Elocon; Drug: Locoid; Other: LEO 90100 foam vehicle
- Dermoval®/Dermovate® (Active Comparator): Dermoval®/Dermovate® (clobetasol propionate 0.05%) cream
  Each subject has all 6 treatments applied topically at the same time, however, the location on which the treatments are applied is randomised. Subjects will receive approximately 20 μl of each investigational product applied in circles with a diameter of 2.2 cm once.
  Interventions: Drug: LEO 90100 aerosol foam; Drug: Dermoval®/Dermovate®; Drug: Diprosone; Drug: Elocon; Drug: Locoid; Other: LEO 90100 foam vehicle
- Diprosone® (Active Comparator): Diprosone® betamethasone 0.5 mg/g (as dipropionate) ointment
  Each subject has all 6 treatments applied topically at the same time, however, the location on which the treatments are applied is randomised. Subjects will receive approximately 20 μl of each investigational product applied in circles with a diameter of 2.2 cm once.
  Interventions: Drug: LEO 90100 aerosol foam; Drug: Dermoval®/Dermovate®; Drug: Diprosone; Drug: Elocon; Drug: Locoid; Other: LEO 90100 foam vehicle
- Elocon® (Active Comparator): Elocon® mometasone furoate 0.1% cream
  Each subject has all 6 treatments applied topically at the same time, however, the location on which the treatments are applied is randomised. Subjects will receive approximately 20 μl of each investigational product applied in circles with a diameter of 2.2 cm once.
  Interventions: Drug: LEO 90100 aerosol foam; Drug: Dermoval®/Dermovate®; Drug: Diprosone; Drug: Elocon; Drug: Locoid; Other: LEO 90100 foam vehicle
- Locoid® (Active Comparator): Locoid® hydrocortisone-17-butyrate 0.1% ointment
  Each subject has all 6 treatments applied topically at the same time, however, the location on which the treatments are applied is randomised. Subjects will receive approximately 20 μl of each investigational product applied in circles with a diameter of 2.2 cm once.
  Interventions: Drug: LEO 90100 aerosol foam; Drug: Dermoval®/Dermovate®; Drug: Diprosone; Drug: Elocon; Drug: Locoid; Other: LEO 90100 foam vehicle
- LEO 90100 foam vehicle (Placebo Comparator): LEO 90100 foam vehicle
  Each subject has all 6 treatments applied topically at the same time, however, the location on which the treatments are applied is randomised. Subjects will receive approximately 20 μl of each investigational product applied in circles with a diameter of 2.2 cm once.
  Interventions: Drug: LEO 90100 aerosol foam; Drug: Dermoval®/Dermovate®; Drug: Diprosone; Drug: Elocon; Drug: Locoid; Other: LEO 90100 foam vehicle

INTERVENTIONS:
Drug: LEO 90100 aerosol foam
Drug: Dermoval®/Dermovate®
Drug: Diprosone
Drug: Elocon
Drug: Locoid
Other: LEO 90100 foam vehicle

SUMMARY:
Vasoconstriction study with LEO 90100

DETAILED DESCRIPTION:
This study compares the pharmacodynamic activity of LEO 90100 with Dermovate cream, Diprosone ointment, Elocon cream, Locoid ointment and LEO 90100 vehicle using a human skin blanching test

ELIGIBILITY:
Inclusion Criteria:

* Subjects demonstrating adequate vasoconstriction to Diprosone® ointment within 15 days prior to dosing (unoccluded application of Diprosone® ointment for 4-6 hours must show a visual score of skin blanching of at least one unit (visual scale (0-4)).
* Subjects without signs of skin irritation/disease/disorders/symptoms or blemishes on test sites (e.g. erythema, dryness, roughness, scaling, scars, moles, sunburn).

Exclusion Criteria:

* Abnormal pigmentation of the skin or skin type that could, in any way, confound interpretation of the trial results (skin type V and VI on the Fitzpatrick scale).
* Female subjects who are breastfeeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Mean of two visual skin blanching scores for each treatment measured 2 hours after 16 hours application under non-occlusive conditions | 18 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CPCAD, Nice, Cedex, France

IPD SHARING:
Plan to Share IPD: No